CLINICAL TRIAL: NCT00344799
Title: Molecular and Cytogenetic Studies of Ocular Melanoma
Brief Title: Cytogenetic Study of Ocular Melanoma
Status: Completed | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UCLA IRB#04-12-084; 11-000847 (Other: University of California at Los Angeles)
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Choroidal Melanoma
Keywords: Choroidal Melanoma; Choroidal Malignant Melanoma; Ocular Melanoma; Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Patients who are diagnosed with choroidal melanoma and undergo I-125 plaque or enucleation surgery consent to participate in the study. A tumor sample taken during surgery is studied in the lab for genetic features. These features and features of subjects' clinical course are recorded. Analysis of the data may identify genetic features that are indicative of prognostic factors including risk of metastasis.

DETAILED DESCRIPTION:
The Jules Stein Eye Institute Ocular Melanoma Research Group is conducting cytogenetic studies of choroidal melanoma to improve the screening of biopsy samples of choroidal melanoma through cytogenetic analysis. Our goal is to identify molecular probes that specifically target regions of chromosomes that undergo changes characteristic of metastatic choroidal melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with diagnosis of ocular melanoma
2. Patient with local treatment plan for ocular melanoma- plaque brachytherapy or enucleation
3. Patient 18 years of age or older
4. Archival enucleation specimens with diagnosis of ocular melanoma

Exclusion Criteria:

1. Patient who refuses local melanoma treatment
2. Patient who refuses to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with ocular melanoma, and underwent melanoma treatment at our facility.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2005-01-08 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara M McCannel, MD, PhD, Principal Investigator — Jules Stein Eye Institute, UCLA; Bradley R Straatsma, MD, JD, Study Director — Jules Stein Eye Institute, UCLA; Lynn Gordon, MD, PhD, Study Chair — Jules Stein Eye Institute, UCLA; Ben Glasgow, MD, Study Chair — Jules Stein Eye Institute, UCLA; Nagesh P Rao, PhD, Study Chair — UCLA Pathology and Laboratory Medicine
Locations (1):
- Jules Stein Eye Institute, Los Angeles, California, United States

REFERENCES:
- [Derived] McCannel TA, Burgess BL, Nelson SF, Eskin A, Straatsma BR. Genomic identification of significant targets in ciliochoroidal melanoma. Invest Ophthalmol Vis Sci. 2011 May 9;52(6):3018-22. doi: 10.1167/iovs.10-5864. PMID 20688739